CLINICAL TRIAL: NCT06440486
Title: Based on a Randomized, Double-blind, Controlled Trial, Evaluate the Effects of Probiotics on Inflammation and Metabolism in Patients With Type 2 Diabetes Mellitus.
Brief Title: Assessment of Probiotics on Inflammation and Metabolism in Type 2 Diabetes.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024008
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Participants will receive a probiotic strip (3g/strip) daily alongside their standard clinical treatment for a continuous 12-week period.
  Interventions: Dietary Supplement: Probiotics
- Maltodextrin (Placebo Comparator): Participants will take a daily placebo strip (3g/strip) in addition to their regular clinical treatment over a continuous 12-week period.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Serum and fecal samples were collected at the beginning and end of the study to evaluate the effects of probiotic consumption on immune markers, metabolites, and gut microbiota before and after administration.

SUMMARY:
This clinical study aims to explore the effects of probiotics on inflammatory and metabolic indicators in patients with type 2 diabetes. By assessing the potential of probiotics to modify these markers, the study seeks to identify an economical and effective strategy for the prevention and treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an informed consent form before the study and has a thorough understanding of the content, process, and possible adverse reactions of the study;
2. Age 18 (inclusive) and above, gender not limited;
3. Diagnosed with type 2 diabetes mellitus;
4. Not diagnosed with cardiovascular, kidney, or any other diabetic complications.

Exclusion Criteria:

1. Age over 75 years old;
2. Use of exogenous insulin or patients with cardiovascular disease and other complications;
3. Patients who are currently using α-glucosidase inhibitors;
4. Patients who have a habit of taking probiotics or are currently taking probiotics;
5. Pregnant or lactating women;
6. Subjects deemed unsuitable for participation in this clinical study by the investigators due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers | 12 weeks
  Blood samples will be collected from patients with type 2 diabetes mellitus (T2DM), centrifuged to obtain serum, and analyzed for tumor necrosis factor-alpha (TNF-α), interleukins 6 (IL-6), 10 (IL-10), and 18 (IL-18), IL-1β, and interferon-gamma (IFN-γ) to assess the impact of probiotics on T2DM patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China

IPD SHARING:
Plan to Share IPD: No